CLINICAL TRIAL: NCT01038089
Title: Pilot Study Of The Effects Of Resveratrol On Endothelial Function In Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Joseph A. Vita, MD, Boston University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-28258
Record Dates: First submitted 2009-12-19; First posted 2009-12-23 (Estimated); Last update posted 2010-12-21 (Estimated); Status verified 2010-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: endothelium; resveratrol; diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Resveratrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- resveratrol (Experimental): Resveratrol
  Interventions: Dietary Supplement: Resveratrol

INTERVENTIONS:
Dietary Supplement: Resveratrol — Resveratrol
  Other Names: ResVida

SUMMARY:
Observational studies have shown that consumption of grapes and grape products such as red wine is associated with reduced cardiovascular risk. The mechanisms accounting for this benefit remain incompletely understood. Resveratrol is a component of grapes and red wine that has favorable effects on endothelial function in diabetic and obese animals. Resveratrol is available to people over-the-counter in health food stores and the internet as a dietary supplement.

The endothelium plays a central role in the control of blood vessel function. When healthy, the endothelium prevents vasospasm, blood clot formation, and the development of atherosclerosis. Endothelial function is abnormal in patients with diabetes mellitus and this abnormality contributes to the development of cardiovascular disease.

The present pilot study is designed to test the hypothesis that resveratrol (90 mg/day and 270 mg/day for one week each) will have favorable effects on endothelial function in patients with diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female subjects.
2. Age over 21 years old.
3. Body mass index greater than or equal to 25 and less than 35 kg/m2
4. Clinically stable Type 2 diabetes mellitus.
5. Willing to give written informed consent and able to understand, to participate in and to comply with the study requirements.
6. Willing to refrain from consumption of red wine, grape juice, and grape products beginning two weeks before and continuing throughout the entire study period.

Exclusion Criteria:

1. Women who lactating or pregnant. All women with childbearing potential will undergo a urine pregnancy test at each visit to exclude pregnancy.
2. Treatment with an investigational product within the last 30 days.
3. Clinically evident major illness of other organ systems, including end-stage cancer, renal failure, or other conditions that in the opinion of the principal investigator make a clinical study inappropriate.
4. Liver transaminase levels greater than 3X the upper limit of normal.
5. History of a psychological illness or condition such as to interfere with the subject's ability to understand the requirements of the study.
6. Vitamin supplements exceeding two times the recommending daily allowance (RDA) within the last 30 days prior to screening.
7. Resveratrol, green tea and isoflavone supplements within the last 30 days prior to screening.
8. Subjects who practice a vegetarian or vegan diet
9. Subjects taking budesonide, buspirone, eplerenone, eletriptan, felodipine, midazolam, saquinavir, sildenafil, triazolam, vardenafil, alfentanil, astemizole, cisapride, cyclosporine, diergotamine, ergotamine, fentanyl, irinotecan, pimozide, quinidine, sirolimus, tacrolimus, terfenadine, or warfarin.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Brachial artery flow-mediated dilation | 2 weeks

SECONDARY OUTCOMES:
Blood markers of inflammation, oxidative stress, insulin resistance | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Vita, MD, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States